CLINICAL TRIAL: NCT00012857
Title: Pain Management and Behavioral Outcomes in Patients With Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NRI 95-192
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Dementia; Alzheimer Disease, Pain; Behavior, Agitation
MeSH Terms: conditions — Dementia; Alzheimer Disease; Pain; Behavior; Psychomotor Agitation | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: acetaminophen 650 mg qid and placebo qid PRN. The other arm was placebo qid and acetaminophen 650 mg qid PRN

INTERVENTIONS:
Drug: acetaminophen 650 mg qid and placebo qid PRN. The other arm was placebo qid and acetaminophen 650 mg qid PRN

SUMMARY:
Dementia illness often co-exists with painful medical conditions associated with aging (e.g., degenerative joint disease, osteoarthritis, skin ulcers, back pain, headaches, cancer, or angina). While the standard practice is pain assessment for all patients, the elderly with dementia have special needs for assessment, management, and evaluation. When they are unable to verbalize pain, objective measurement of their discomfort are possible manifestations of pain. No research relates systemic pain treatment with reduction of negative problematic behaviors in patient dementia.

DETAILED DESCRIPTION:
Background:

Dementia illness often co-exists with painful medical conditions associated with aging (e.g., degenerative joint disease, osteoarthritis, skin ulcers, back pain, headaches, cancer, or angina). While the standard practice is pain assessment for all patients, the elderly with dementia have special needs for assessment, management, and evaluation. When they are unable to verbalize pain, objective measurement of their discomfort are possible manifestations of pain. No research relates systemic pain treatment with reduction of negative problematic behaviors in patient dementia.

Objectives:

The objectives of this research are (1) to elucidate the relationships between pain, discomfort, and agitation; and (2) to determine the influence that pain management has on decreasing the outcomes of discomfort, agitation, and confusion in nursing home residents.

Methods:

This study used a randomized, double-blind, placebo-controlled, cross-over design. Each treatment arm lasted two weeks. The crossover point occurred without washout. One arm was acetaminophen 650 mg qid and placebo qid PRN. The other arm was placebo qid and acetaminophen 650 mg qid PRN. Sites involved in the study included the Jewish Home for the Aged in San Francisco; Golden Gate Healthcare Center in San Francisco; Palo Alto VA Health Care System; Nursing Home Care Unit at Livermore. Patients were included who: are > 55 years; have severe dementia; have a documented painful condition not requiring opiates or a current medication regimen; unable to report pain consistently or reliably; be present and accept treatment for study duration; have > 1 episode of agitation per day. Patients with schizophrenia or severe Parkinson�s are excluded. A research assistant (blind to treatment arm) tested each patient for discomfort, agitation, and confusion at baseline and two times per day on two days of the week for four weeks. Nurses rated patients for agitation each shift. Instruments included the Cohen-Mansfield Agitation Inventory, the Discomfort Scale, and the Confusion Assessment Method. Repeated measures analyses examined effect of treatment on the three behaviors (agitation, confusion, and discomfort).

Status:

The study is complete. Final report was submitted to HSR&D in August 2001.

ELIGIBILITY:
Inclusion Criteria:

Patients must be: 55 years old and older, nursing home residents, a diagnosed painful that would respond to tylenol, documented agitated behavior, a dementia diagnosis or a functional impairment severe enough to rate a 7 on the Global Deterioration Scale, be unable to report pain. Patients must have been residents in the nursing home for at least 1 month with a plan to stay at least 2 months.

Exclusion Criteria:

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn K. Douglas, DNSc RN FAAN, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States